CLINICAL TRIAL: NCT00882388
Title: Phase 4 Study of the Effect of Celecoxib on the Antiplatelet Effect of Aspirin and Clopidogrel
Brief Title: The Effect of Celecoxib on the Antiplatelet Effect of Aspirin and Clopidogrel in Normal Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyo-Soo Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COREA-volunteer
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: celecoxib; platelet; thrombosis; Volunteers
MeSH Terms: conditions — Thrombosis | interventions — Aspirin; Celecoxib; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ASA (Active Comparator): aspirin only
  Interventions: Drug: aspirin
- Cele (Active Comparator)
  Interventions: Drug: celecoxib
- ASA + Cele (Experimental)
  Interventions: Drug: aspirin + celecoxib
- ASA + Clo (Active Comparator)
  Interventions: Drug: aspirin + clopidogrel
- ASA + Clo + Cele (Experimental)
  Interventions: Drug: aspirin + clopidogrel + celecoxib

INTERVENTIONS:
Drug: aspirin — aspirin 100 mg qd for 7 days
  Other Names: aspirin : Keun-Hwa Phamaceutical; clopidogrel : sanofi-aventis; celecoxib : Pfizer
  Arms: ASA
Drug: celecoxib — celecoxib 200 mg bid * 7 days
  Other Names: aspirin : Keun-Hwa Phamaceutical; clopidogrel : sanofi-aventis; celecoxib : Pfizer
  Arms: Cele
Drug: aspirin + celecoxib — aspirin 100 mg qd + celecoxib 200 mg bid for 7 days
  Other Names: aspirin : Keun-Hwa Phamaceutical; clopidogrel : sanofi-aventis; celecoxib : Pfizer
  Arms: ASA + Cele
Drug: aspirin + clopidogrel — asprin 100 mg qd + clopidogrel 75 mg qd for 7 days
  Other Names: aspirin : Keun-Hwa Phamaceutical; clopidogrel : sanofi-aventis; celecoxib : Pfizer
  Arms: ASA + Clo
Drug: aspirin + clopidogrel + celecoxib — aspirin 100 mg qd + clopidogrel 75 mg qd + celecoxib 200 mg bid
  Other Names: aspirin : Keun-Hwa Phamaceutical; clopidogrel : sanofi-aventis; celecoxib : Pfizer
  Arms: ASA + Clo + Cele

SUMMARY:
Background:

* The prevalence of arthritis which needs celecoxib prescription is high in patients with coronary artery disease.
* The main concern is that celecoxib would increase thrombogenicity by inhibiting the synthesis of prostacyclin in endothelial cells.
* It is not known whether the administration of celecoxib would deteriorate antiplatelet effects of aspirin and clopidogrel which are used after stenting.

Methods:

* Healthy volunteers (n=40)
* Randomization into five subgroups
* aspirin, celecoxib, aspirin+celecoxib, aspirin+clopidogrel, aspirin+clopidogrel+celecoxib
* Medication schedule : medication of each drug for 6 days, blood samples at day 0 and day 7
* Celecoxib 200mg twice a day, and/or aspirin 100mg daily, and/or clopidogrel 75 mg daily
* Platelet function test : light transmittance aggregometry and arachidonic acid metabolite assay among subgroups.

Study hypothesis : The addition of celecoxib does not deteriorate antiplatelet function of aspirin and clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers including both men and women 20~30 years
* no abnormality in physical examination, 12-lead ECG, and routine laboratory test

Exclusion Criteria:

* Subjects with cardiovascular disease, hemostatic disorder, hypersensitivity to NSAIDs and clopidogrel
* Women with a positive pregnancy test
* smoker
* chronic drinkers
* overweight exceeding 20% of standard body weight

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Light transmittance aggregometry : % of inhibition (ADP, collagen) | 7 days

SECONDARY OUTCOMES:
Urine arachidonic metabolite assay | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea